CLINICAL TRIAL: NCT04441008
Title: Radical aiTBS Protocol for Intractable Depression
Brief Title: Accelerated iTBS for Depression and Suicidality
Acronym: RAPID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Nicholas Trapp, Assistant Professor of Psychiatry, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202002608
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder; Suicide
Keywords: transcranial magnetic stimulation, theta burst, accelerated TMS, ECT, electroconvulsive therapy, depression, suicidality
MeSH Terms: conditions — Depressive Disorder, Major; Suicide; Epilepsy, Rolandic; Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Single-blind with crossover of experimental (aiTBS) group into standard of care (ECT) group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor will be blinded to patient's designation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- aiTBS arm (Experimental): aiTBS treatment as lead-in phase to ECT standard of care treatment.
  Interventions: Device: Accelerated Intermittent Theta Burst (aiTBS); Device: Electroconvulsive therapy (ECT)
- ECT arm (Active Comparator): ECT as clinically indicated.
  Interventions: Device: Electroconvulsive therapy (ECT)

INTERVENTIONS:
Device: Accelerated Intermittent Theta Burst (aiTBS) — High-dose intermittent theta burst administered at a treatment frequency 10x per day, with each treatment session duration 3x standard TMS (1800 pulses). Delivering 50 sessions in 5 days.
  Other Names: SAINT Protocol, accelerated TMS
  Arms: aiTBS arm
Device: Electroconvulsive therapy (ECT) — ECT as per standard clinical care and management.

SUMMARY:
The overall objective of this current study is to evaluate the feasibility, safety, and tolerability of "high dose" aiTBS in psychiatric inpatient and outpatients with treatment-refractory unipolar, non-psychotic major depressive disorder, using patients receiving ECT as an active comparator. Developing a better understanding of the feasibility and tolerability of adapting this treatment to an acutely ill patient population could lead to huge breakthroughs for clinician decision-making and for the further optimization of brain stimulation depression protocols. The results of this study can help guide future confirmatory efficacy trials of high-dose aiTBS by providing a better understanding of how feasibility, safety and tolerability compare to ECT, as well as unforeseen challenges of its use.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to provide informed consent

  * Availability for the duration of the study and willingness to comply with all study procedures
  * Age 18 to 90
  * Diagnosis of major depressive disorder by DSM-5 criteria
  * Depressive symptoms are thought to be caused primarily by a major depressive episode and not by some other neurologic or psychiatric illness
  * Failure of or intolerance to at least 2 antidepressant treatments of different therapeutic classes (can include psychotherapy trial or neurostimulation trial)
  * Meets criteria for clinical eligibility for ECT treatment, including optimization of any medical conditions and completion of any medical testing or clearance as clinically indicated
  * Able to consent voluntarily to treatment
  * Score of at least 2 on the MADRS item 10
  * Ability to sit or lie down for an extended period of time and willingness to adhere to the theta burst stimulation protocol

Exclusion Criteria:

* • Presence of implanted ferromagnetic devices or materials, including cardiac pacemaker, cochlear implant, deep brain stimulation device, vagus nerve stimulation device, shrapnel, facial or scalp piercings that cannot be removed, or metallic face or head tattoos

  * Pregnancy or lactation
  * Previous bad reaction or intolerance to transcranial magnetic stimulation
  * Febrile illness within 1 week
  * Treatment with another investigational drug or other intervention within 30 days
  * Recent substance abuse or use disorder within the past 6 months, excluding tobacco or infrequent cannabis use
  * History of epilepsy or seizure disorder
  * History of penetrating traumatic brain injury, multiple sclerosis, or history of brain surgery or intracranial hemorrhage
  * Primary psychiatric or medical/neurologic illness other than MDD that is more likely to account for depressive symptoms, including severe personality disorder or psychotic illness
  * Severe or moderate intellectual disability
  * Major neurocognitive disorder
  * Involuntary commitment or petition filed for involuntary ECT treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Retention rate at completion of aiTBS vs the ECT group | 5 days
  The primary tolerability endpoint is the proportion of aiTBS or ECT patients completing the protocol to a degree thought to be satisfactory for achieving the intended antidepressant effect. Completion for aiTBS arm is defined as completion of at least 60% of the treatment protocol (30 of 50 treatments) with treatments on at least 60% of days (3 of 5 days during the week). Completion for ECT arm is defined as completion of at least 2 of 3 ECT treatments during the first week.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Trapp, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perera T, George MS, Grammer G, Janicak PG, Pascual-Leone A, Wirecki TS. The Clinical TMS Society Consensus Review and Treatment Recommendations for TMS Therapy for Major Depressive Disorder. Brain Stimul. 2016 May-Jun;9(3):336-346. doi: 10.1016/j.brs.2016.03.010. Epub 2016 Mar 16. PMID 27090022
- [Background] Levkovitz Y, Isserles M, Padberg F, Lisanby SH, Bystritsky A, Xia G, Tendler A, Daskalakis ZJ, Winston JL, Dannon P, Hafez HM, Reti IM, Morales OG, Schlaepfer TE, Hollander E, Berman JA, Husain MM, Sofer U, Stein A, Adler S, Deutsch L, Deutsch F, Roth Y, George MS, Zangen A. Efficacy and safety of deep transcranial magnetic stimulation for major depression: a prospective multicenter randomized controlled trial. World Psychiatry. 2015 Feb;14(1):64-73. doi: 10.1002/wps.20199. PMID 25655160
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Peng Z, Zhou C, Xue S, Bai J, Yu S, Li X, Wang H, Tan Q. Mechanism of Repetitive Transcranial Magnetic Stimulation for Depression. Shanghai Arch Psychiatry. 2018 Apr 25;30(2):84-92. doi: 10.11919/j.issn.1002-0829.217047. PMID 29736128
- [Background] Williams NR, Sudheimer KD, Bentzley BS, Pannu J, Stimpson KH, Duvio D, Cherian K, Hawkins J, Scherrer KH, Vyssoki B, DeSouza D, Raj KS, Keller J, Schatzberg AF. High-dose spaced theta-burst TMS as a rapid-acting antidepressant in highly refractory depression. Brain. 2018 Mar 1;141(3):e18. doi: 10.1093/brain/awx379. No abstract available. PMID 29415152
- [Background] Friedrich MJ. Depression Is the Leading Cause of Disability Around the World. JAMA. 2017 Apr 18;317(15):1517. doi: 10.1001/jama.2017.3826. No abstract available. PMID 28418490
- [Background] Zhan Y, Zhang B, Zhou Y, Zheng W, Liu W, Wang C, Li H, Chen L, Yu L, Walter M, Li M, Li MD, Ning Y. A preliminary study of anti-suicidal efficacy of repeated ketamine infusions in depression with suicidal ideation. J Affect Disord. 2019 May 15;251:205-212. doi: 10.1016/j.jad.2019.03.071. Epub 2019 Mar 22. PMID 30927581
- [Background] Baeken C. Accelerated rTMS: A Potential Treatment to Alleviate Refractory Depression. Front Psychol. 2018 Oct 31;9:2017. doi: 10.3389/fpsyg.2018.02017. eCollection 2018. PMID 30429807
- [Background] Feffer K, Lee HH, Mansouri F, Giacobbe P, Vila-Rodriguez F, Kennedy SH, Daskalakis ZJ, Blumberger DM, Downar J. Early symptom improvement at 10 sessions as a predictor of rTMS treatment outcome in major depression. Brain Stimul. 2018 Jan-Feb;11(1):181-189. doi: 10.1016/j.brs.2017.10.010. Epub 2017 Oct 19. PMID 29107623
- [Background] Hawley CJ, Gale TM, Sivakumaran T; Hertfordshire Neuroscience Research group. Defining remission by cut off score on the MADRS: selecting the optimal value. J Affect Disord. 2002 Nov;72(2):177-84. doi: 10.1016/s0165-0327(01)00451-7. PMID 12200208
- [Background] Kerner N, Prudic J. Current electroconvulsive therapy practice and research in the geriatric population. Neuropsychiatry (London). 2014 Feb;4(1):33-54. doi: 10.2217/npy.14.3. PMID 24778709
- [Background] Guse B, Falkai P, Wobrock T. Cognitive effects of high-frequency repetitive transcranial magnetic stimulation: a systematic review. J Neural Transm (Vienna). 2010 Jan;117(1):105-22. doi: 10.1007/s00702-009-0333-7. Epub 2009 Oct 27. PMID 19859782
- [Background] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434